CLINICAL TRIAL: NCT03658629
Title: Phase 2 Clinical Trial to Confirm the Dose and Formulation of a Recombinant Quadrivalent Nanoparticle Influenza Vaccine (Quad-NIV) With or Without Matrix-M1™ Adjuvant in Healthy Adults ≥ 65 Years of Age
Brief Title: Phase 2 Dose and Formulation Confirmation of Quad-NIV in Older Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated 182 days after initial dosing.
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: qNIV-E-201
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose A (Experimental): Alternating deltoid injections of Quad-NIV (60 µg HA per A strain and B strain; in-clinic mix with 50 µg of Matrix-M1) on Day 0 and Placebo on Day 28.
  Interventions: Biological: NanoFlu (Quad-NIV); Other: Matrix-M Adjuvant; Other: Placebo
- Dose B (Experimental): Alternating deltoid injections of Quad-NIV (60 µg HA per A strain and B strain; co-formulated with 50 µg of Matrix-M1) on Day 0 and Placebo on Day 28.
  Interventions: Biological: NanoFlu (Quad-NIV); Other: Matrix-M Adjuvant; Other: Placebo
- Dose C (Experimental): Alternating deltoid injections of Quad-NIV (60 µg HA per A strain and B strain; co-formulated with 75 µg of Matrix-M1) on Day 0 and Placebo on Day 28.
  Interventions: Biological: NanoFlu (Quad-NIV); Other: Matrix-M Adjuvant; Other: Placebo
- Dose D (Experimental): Alternating deltoid injections of Quad-NIV (60 µg HA per A strain and 90 µg HA per B strain; co-formulated with 50 µg of Matrix-M1) on Day 0 and Placebo on Day 28.
  Interventions: Biological: NanoFlu (Quad-NIV); Other: Matrix-M Adjuvant; Other: Placebo
- Dose E (Experimental): Alternating deltoid injections of Quad-NIV (60 µg HA per A and B strain without adjuvant) on Day 0 and Licensed 2018-2019 Influenza vaccine on Day 28.
  Interventions: Biological: NanoFlu (Quad-NIV); Biological: Influenza Vaccine
- Dose F (Experimental): Alternating deltoid injections of 2018-2019 High-Dose Trivalent Vaccine on Day 0 and Placebo on Day 28.
  Interventions: Other: Placebo; Biological: Fluzone HD
- Dose G (Experimental): Alternating deltoid injections of 2018-2019 Quadrivalent Vaccine on Day 0 and Placebo on Day 28.
  Interventions: Other: Placebo; Biological: Flublok Quadrivalent

INTERVENTIONS:
Biological: NanoFlu (Quad-NIV) — 2018-2019 Investigational Quadrivalent Seasonal Influenza Vaccine
  Arms: Dose A; Dose B; Dose C; Dose D; Dose E
Other: Matrix-M Adjuvant — Adjuvant
  Arms: Dose A; Dose B; Dose C; Dose D
Other: Placebo — Placebo
  Arms: Dose A; Dose B; Dose C; Dose D; Dose F; Dose G
Biological: Fluzone HD — 2018-2019 Licensed Trivalent Seasonal Influenza Vaccine
  Arms: Dose F
Biological: Flublok Quadrivalent — 2018-2019 Licensed Quadrivalent Seasonal Influenza Vaccine
  Arms: Dose G
Biological: Influenza Vaccine — 2018-19 Licensed Seasonal Influenza Vaccine
  Arms: Dose E

SUMMARY:
A Phase 2 trial to confirm the dose and formulation, demonstrate adjuvant effect, and evaluate the safety and tolerability of a single intramuscular injection of Quad-NIV with or without Matrix-M1 adjuvant in healthy adults ≥ 65 years of age.

A total of approximately 1375 subjects were to be randomized to seven treatment groups to receive Quad-NIV or an active comparator.

DETAILED DESCRIPTION:
This randomized, observer-blind, active-controlled, Phase 2 trial was conducted at multiple sites. The composition of the Quad-NIV Influenza Vaccines used in this trial included recombinant H1, H3, and two B hemagglutinin proteins for the 2018-2019 Northern Hemisphere influenza virus strains.

Approximately 1375 healthy male and female subjects ≥ 65 years were randomized into 7 treatment groups (group A to group G), receiving various formulations of Quad-NIV, with or without Matrix-M1 adjuvant or one of two active comparator influenza vaccines. Within each site, randomization was stratified by history of receipt of 2017-2018 influenza vaccine. Subjects received two injections 28 days apart. On Day 0, subjects received one of the five Quad-NIV formulations or one of the two comparator influenza vaccines. On Day 28, subjects received either placebo or a licensed influenza vaccine rescue dose, depending on his or her initial randomization.

Subjects were followed for safety for approximately 6 months, with primary immunogenicity results at Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically-stable adult male or female, ≥ 65 years of age. Subjects may have 1 or more chronic medical diagnoses, but should be clinically stable as assessed by:

   * Absence of changes in medical therapy within 1 month due to treatment failure or toxicity,
   * Absence of medical events qualifying as serious adverse events within 2 months; and
   * Absence of known, current, and life-limiting diagnoses which render survival to completion of the protocol unlikely in the opinion of the investigator.
2. Willing and able to give informed consent prior to trial enrollment, and
3. Living in the community and able to attend trial visits, comply with trial requirements, and provide timely, reliable, and complete reports of adverse events.

Exclusion Criteria:

1. Participation in research involving investigational product (drug / biologic / device) within 45 days before planned date of first injection.
2. Participation in any previous Novavax's influenza vaccine clinical trial(s).
3. History of a serious reaction to prior influenza vaccination, known allergy to constituents of licensed comparator vaccines or polysorbate 80.
4. History of Guillain-Barré Syndrome (GBS) within 6 weeks following a previous influenza vaccine.
5. Received any vaccine in the 4 weeks preceding the trial vaccination and any influenza vaccine within 6 months preceding the trial vaccination.
6. Any known or suspected immunosuppressive illness, congenital or acquired, based on medical history and/or physical examination.
7. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the trial vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
8. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the trial vaccine or during the trial.
9. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature ≥ 38.0°C, on the planned day of vaccine administration).
10. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of trial results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
11. Known disturbance of coagulation.
12. Suspicion or recent history (within 1 year of planned vaccination) of alcohol or other substance abuse.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1375 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax
Locations (14):
- United States (14):
  - US135, Hollywood, Florida
  - US045, Savannah, Georgia
  - US013, Stockbridge, Georgia
  - US138, Rockville, Maryland
  - US025, Norfolk, Nebraska
  - US018, Omaha, Nebraska
  - US078, Cary, North Carolina
  - US108, Raleigh, North Carolina
  - US137, Salisbury, North Carolina
  - US132, Statesville, North Carolina
  - US071, Wilmington, North Carolina
  - US063, Winston-Salem, North Carolina
  - US056, Moncks Corner, South Carolina
  - US050, Dakota Dunes, South Dakota

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shinde V, Cai R, Plested J, Cho I, Fiske J, Pham X, Zhu M, Cloney-Clark S, Wang N, Zhou H, Zhou B, Patel N, Massare MJ, Fix A, Spindler M, Thomas DN, Smith G, Fries L, Glenn GM. Induction of Cross-Reactive Hemagglutination Inhibiting Antibody and Polyfunctional CD4+ T-Cell Responses by a Recombinant Matrix-M-Adjuvanted Hemagglutinin Nanoparticle Influenza Vaccine. Clin Infect Dis. 2021 Dec 6;73(11):e4278-e4287. doi: 10.1093/cid/ciaa1673. PMID 33146720
- See also: Related Info — http://novavax.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Alternating deltoid injections of Quad-NIV (60 µg HA per A strain and B strain; in-clinic mix with 50 µg of Matrix-M1) on Day 0 and Placebo on Day 28.
- Group B: Alternating deltoid injections of Quad-NIV (60 µg HA per A strain and B strain; co-formulated with 50 µg of Matrix-M1) on Day 0 and Placebo on Day 28.
- Group C: Alternating deltoid injections of Quad-NIV (60 µg HA per A strain and B strain; co-formulated with 75 µg of Matrix-M1) on Day 0 and Placebo on Day 28.
- Group D: Alternating deltoid injections of Quad-NIV (60 µg HA per A strain and 90 µg HA per B strain; co-formulated with 50 µg of Matrix-M1) on Day 0 and Placebo on Day 28.
- Group E: Alternating deltoid injections of Quad-NIV (60 µg HA per A and B strain without adjuvant) on Day 0 and Licensed 2018-2019 Influenza vaccine on Day 28.
- Group F: Alternating deltoid injections of 2018-2019 High-Dose Trivalent Vaccine on Day 0 and Placebo on Day 28.
- Group G: Alternating deltoid injections of 2018-2019 Quadrivalent Vaccine on Day 0 and Placebo on Day 28.
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Group G
Started | 158 | 309 | 155 | 133 | 313 | 154 | 153
Participants in Safety Population | 157 | 305 | 156 | 132 | 311 | 153 | 151
Completed | 151 | 296 | 149 | 125 | 303 | 151 | 148
Not Completed | 7 | 13 | 6 | 8 | 10 | 3 | 5

BASELINE CHARACTERISTICS:
Population: The population analyzed is the number of participants that are in the Safety Population.
Groups:
- Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A: Alternating deltoid injections of 2018-2019 Quad-NIV-1 (Day 0) and Placebo (Day 28)
  NanoFlu (Quad-NIV): 2018-2019 Investigational Quadrivalent Seasonal Influenza Vaccine
  Matrix-M Adjuvant: Adjuvant
  Placebo: Placebo
- Quad-NIV Preformulated With Adjuvant Dose A: Alternating deltoid injections of 2018-2019 Quad-NIV-2 (Day 0) and Placebo (Day 28)
  NanoFlu (Quad-NIV): 2018-2019 Investigational Quadrivalent Seasonal Influenza Vaccine
  Matrix-M Adjuvant: Adjuvant
  Placebo: Placebo
- Quad-NIV Preformulated With Adjuvant Dose B: Alternating deltoid injections of 2018-2019 Quad-NIV-3 (Day 0) and Placebo (Day 28)
  NanoFlu (Quad-NIV): 2018-2019 Investigational Quadrivalent Seasonal Influenza Vaccine
  Matrix-M Adjuvant: Adjuvant
  Placebo: Placebo
- Quad-NIV Preformulated With Increased B HA Adjuvant Dose A: Alternating deltoid injections of 2018-2019 Quad-NIV-4 (Day 0) and Placebo (Day 28)
  NanoFlu (Quad-NIV): 2018-2019 Investigational Quadrivalent Seasonal Influenza Vaccine
  Matrix-M Adjuvant: Adjuvant
  Placebo: Placebo
- Quad-NIV Without Adjuvant: Alternating deltoid injections of 2018-2019 Quad-NIV-5 (Day 0) and Licensed 2018-2019 Influenza vaccine (Day 28)
  NanoFlu (Quad-NIV): 2018-2019 Investigational Quadrivalent Seasonal Influenza Vaccine
  Fluzone HD: 2018-2019 Licensed Trivalent Seasonal Influenza Vaccine
  Flublok Quadrivalent: 2018-2019 Licensed Quadrivalent Seasonal Influenza Vaccine
- Licensed High-Dose Trivalent Influenza Vaccine: Alternating deltoid injections of 2018-2019 High-Dose Trivalent Vaccine (Day 0) and Placebo (Day 28)
  Placebo: Placebo
  Fluzone HD: 2018-2019 Licensed Trivalent Seasonal Influenza Vaccine
- Licensed Quadrivalent Influenza Vaccine: Alternating deltoid injections of 2018-2019 Quadrivalent Vaccine (Day 0) and Placebo (Day 28)
  Placebo: Placebo
  Flublok Quadrivalent: 2018-2019 Licensed Quadrivalent Seasonal Influenza Vaccine
- Total: Total of all reporting groups
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine | Total
Number analyzed (Participants) | 157 | 305 | 156 | 132 | 311 | 153 | 151 | 1365
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (5.5) | 72.0 (5.5) | 71.8 (5.6) | 72.6 (6.1) | 72.6 (6.3) | 72.5 (5.5) | 72.9 (5.6) | 72.7 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Population analyzed is the number of participants that completed the study. Safety Population
  Participants
    Female | 90 | 179 | 77 | 81 | 185 | 99 | 87 | 798
    Male | 67 | 126 | 79 | 51 | 126 | 54 | 64 | 567
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 7 | 4 | 7 | 6 | 4 | 40
  Not Hispanic or Latino | 151 | 299 | 149 | 128 | 304 | 147 | 147 | 1325
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Population analyzed is the number of participants that completed the study. Safety Population
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 5
    Asian | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Black or African American | 13 | 41 | 15 | 12 | 29 | 17 | 14 | 141
    White | 138 | 261 | 140 | 120 | 277 | 133 | 135 | 1204
    More than one race | 3 | 1 | 1 | 0 | 1 | 2 | 0 | 8
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs)
Description: Adverse Events over the 7 days post-injection; all adverse events (including adverse changes in clinical laboratory parameters) through 21 days post-injection; and Medically Attended Adverse Events (MAEs), Serious Adverse Events (SAEs), and Significant New Medical Conditions (SNMCs) through 6 months post-injection.
Time Frame: Day 0 - Day 182
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 157 | 305 | 156 | 132 | 311 | 153 | 151
participants
  All AE's | 100 | 189 | 92 | 71 | 165 | 93 | 87
  SAE's | 8 | 16 | 8 | 12 | 6 | 6 | 3
  MAE's | 51 | 87 | 29 | 38 | 74 | 34 | 40
  SNMC's | 5 | 18 | 10 | 10 | 15 | 6 | 9

2. Primary Outcome: Hemagglutination Inhibition (HAI) Titers Specific for Vaccine Homologous A and B Influenza Strains Expressed as Geometric Man Titer (GMT)
Description: HAI antibody titers specific for the HA receptor binding domains of vaccine homologous A and B strain(s) at Days 0 and Day 28 post-vaccination expressed as geometric man titer (GMT).
Time Frame: Day 0 - Day 28
Population: Per-Protocol Population for immunogenicity was used for the primary outcome measure and included all randomized subjects that received the assigned dose of the test article according to protocol, had HAI serology results for Day 0 and Day 28, and had no major protocol deviations affecting the primary immunogenicity outcomes.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 149 | 295 | 147 | 121 | 290 | 143 | 144
titers
  Day 0 (A/Michigan/45/2015 (H1N1)) | 50.1 [44.6 to 56.4] | 47.9 [44.2 to 51.9] | 55.3 [49.0 to 62.3] | 48.7 [42.6 to 55.8] | 48.7 [44.8 to 52.8] | 50.5 [45.2 to 56.4] | 44.0 [39.5 to 49.1]
  Day 28 (A/Michigan/45/2015 (H1N1)) | 98.9 [86.4 to 113.1] | 91.3 [82.5 to 101.0] | 99.1 [86.2 to 114.0] | 79.5 [68.6 to 92.2] | 90.3 [81.0 to 100.5] | 96.9 [84.5 to 111.1] | 82.1 [71.6 to 94.2]
  Day 0 (B/Colorado/06/2017 (Victoria Lineage)) | 47.6 [43.1 to 52.6] | 46.4 [42.8 to 50.2] | 48.5 [44.0 to 53.6] | 52.7 [46.7 to 59.4] | 47.5 [43.9 to 51.3] | 52.0 [46.1 to 58.5] | 42.9 [38.5 to 47.7]
  Day 28 (B/Colorado/06/2017 (Victoria Lineage)) | 86.8 [77.1 to 97.7] | 83.2 [76.0 to 91.0] | 89.6 [79.3 to 101.2] | 95.5 [82.2 to 110.3] | 73.2 [67.6 to 79.3] | 93.2 [81.6 to 106.5] | 83.3 [73.2 to 94.9]
  Day 0 (B/Phuket/3073/2013 (Yamagata Lineage)) | 50.4 [44.7 to 56.7] | 47.7 [44.4 to 51.3] | 47.6 [42.9 to 52.9] | 53.6 [46.9 to 61.2] | 48.8 [45.2 to 52.7] | 52.9 [47.3 to 59.1] | 46.9 [42.1 to 52.2]
  Day 28 (B/Phuket/3073/2013 (Yamagata Lineage)) | 108.5 [96.2 to 122.4] | 101.7 [93.3 to 110.3] | 104.9 [92.4 to 119.2] | 113.8 [97.6 to 132.6] | 87.5 [79.5 to 96.4] | 64.5 [57.3 to 72.6] | 102.0 [88.6 to 117.4]
  Day 0 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 21.4 [18.9 to 24.3] | 22.0 [20.0 to 24.1] | 22.8 [19.7 to 26.3] | 23.4 [20.2 to 27.1] | 21.3 [19.3 to 23.5] | 23.2 [20.4 to 26.4] | 19.5 [17.1 to 22.2]
  Day 28 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 65.8 [55.2 to 78.4] | 65.4 [58.3 to 73.5] | 64.2 [54.2 to 76.2] | 59.4 [50.0 to 70.5] | 50.8 [45.0 to 57.4] | 46.5 [38.6 to 55.9] | 66.6 [54.9 to 80.9]

3. Primary Outcome: HAI Titers Specific for Antigenically-drifted Influenza Strains Expressed as GMT
Description: HAI antibody titers specific for at least 2 antigenically-drifted influenza strains, at Days 0 and 28 post-vaccination expressed as geometric man titer (GMT).
Time Frame: Day 0 - Day 28
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 149 | 295 | 147 | 121 | 290 | 143 | 144
titers
  Day 0 (A/Switzerland/9715293/2013 (H3N2))) | 54.6 [47.8 to 62.4] | 60.0 [54.3 to 66.2] | 60.9 [52.7 to 70.3] | 60.6 [52.1 to 70.5] | 58.6 [52.8 to 65.1] | 62.3 [54.3 to 71.6] | 54.8 [47.8 to 62.9]
  Day 28 (A/Switzerland/9715293/2013 (H3N2)) | 146.8 [124.0 to 173.9] | 160.4 [143.9 to 178.7] | 154.8 [132.7 to 180.7] | 137.9 [117.2 to 162.2] | 122.4 [109.1 to 137.3] | 133.4 [111.2 to 160.0] | 158.8 [132.2 to 190.9]
  Day 0 (A/Wisconsin/19/2017 (H3N2)) | 21.7 [19.2 to 24.6] | 23.1 [21.1 to 25.3] | 24.0 [20.7 to 27.7] | 23.9 [20.9 to 27.3] | 22.1 [20.1 to 24.4] | 24.5 [21.6 to 27.7] | 20.7 [18.1 to 23.6]
  Day 28 (A/Wisconsin/19/2017 (H3N2)) | 61.1 [51.8 to 72.0] | 63.2 [56.3 to 70.9] | 63.0 [53.5 to 74.2] | 58.2 [48.9 to 69.2] | 50.1 [44.4 to 56.5] | 46.1 [38.7 to 55.1] | 64.3 [53.5 to 77.2]

4. Secondary Outcome: HAI Titers Specific for Vaccine-homologous A and B Influenza Strains Expressed as GMT
Description: HAI antibody titers specific for the HA receptor binding domains of vaccine-homologous A and B strain(s) expressed as GMT on Day 0,28,56 and 182.
Time Frame: Day 0 - Day 182
Population: Per-Protocol Population for immunogenicity was used for this display of secondary outcome measures and included all randomized subjects that received the assigned dose of the test article according to protocol, had HAI serology results for Day 0 and Day 28, and had no major protocol deviations affecting the primary immunogenicity outcomes
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 149 | 295 | 147 | 121 | 290 | 143 | 144
titers
  Day 0 (A/Michigan/45/2015 (H1N1)) | 45.7 [40.2 to 51.9] | 45.6 [41.8 to 49.8] | 48.3 [42.3 to 55.2] | 43.1 [37.6 to 49.4] | 46.3 [42.4 to 50.5] | 48.3 [42.4 to 55.1] | 40.8 [36.7 to 45.3]
  Day 28 (A/Michigan/45/2015 (H1N1)) | 86.4 [74.4 to 100.3] | 78.9 [70.8 to 87.9] | 84.5 [72.3 to 98.7] | 66.2 [56.6 to 77.5] | 80.3 [72.0 to 89.6] | 92.7 [79.6 to 108.1] | 74.2 [64.2 to 85.9]
  Day 56 (A/Michigan/45/2015 (H1N1)) | 71.0 [61.2 to 82.5] | 62.8 [56.7 to 69.7] | 68.2 [58.5 to 79.7] | 52.7 [45.5 to 61.2] | 81.4 [73.0 to 90.8] | 72.4 [63.0 to 83.2] | 57.1 [49.8 to 65.5]
  Day 182 (A/Michigan/45/2015 (H1N1)) | 62.0 [53.4 to 72.0] | 55.5 [50.3 to 61.3] | 63.1 [54.2 to 73.6] | 50.4 [43.7 to 58.1] | 66.8 [60.4 to 73.8] | 67.0 [58.9 to 76.2] | 50.6 [44.2 to 58.0]
  Day 0 (B/Colorado/06/2017 (Victoria Lineage)) | 99.8 [88.5 to 112.5] | 90.4 [82.7 to 98.9] | 95.0 [83.8 to 107.8] | 108.1 [93.3 to 125.1] | 100.2 [91.9 to 109.1] | 99.5 [87.9 to 112.6] | 88.7 [79.2 to 99.3]
  Day 28 (B/Colorado/06/2017 (Victoria Lineage)) | 159.3 [138.9 to 182.6] | 142.1 [128.0 to 157.8] | 154.8 [133.9 to 179.0] | 173.9 [149.0 to 202.9] | 135.8 [124.1 to 148.7] | 184.1 [159.7 to 212.3] | 141.9 [123.7 to 162.7]
  Day 56 (B/Colorado/06/2017 (Victoria Lineage)) | 132.6 [115.7 to 152.0] | 122.5 [110.4 to 135.9] | 134.0 [116.4 to 154.3] | 147.3 [124.8 to 173.9] | 156.0 [143.0 to 170.1] | 156.4 [134.2 to 182.2] | 113.4 [98.7 to 130.3]
  Day 128 (B/Colorado/06/2017 (Victoria Lineage)) | 119.6 [103.8 to 137.8] | 107.2 [96.2 to 119.2] | 122.1 [105.3 to 141.6] | 131.8 [112.5 to 154.3] | 141.4 [128.4 to 155.7] | 141.9 [123.6 to 162.9] | 108.5 [93.8 to 125.5]
  Day 0 (B/Phuket/3073/2013 (Yamagata Lineage)) | 104.0 [92.0 to 117.7] | 97.1 [89.4 to 105.5] | 94.1 [84.1 to 105.3] | 105.0 [90.5 to 121.9] | 99.7 [91.9 to 108.1] | 100.0 [88.6 to 112.8] | 85.4 [77.0 to 94.6]
  Day 28 (B/Phuket/3073/2013 (Yamagata Lineage)) | 202.4 [175.8 to 233.0] | 195.6 [177.1 to 216.0] | 205.9 [180.1 to 235.4] | 211.2 [178.0 to 250.7] | 179.5 [162.3 to 198.4] | 137.0 [120.6 to 155.6] | 174.9 [150.7 to 203.0]
  Day 56 (B/Phuket/3073/2013 (Yamagata Lineage)) | 192.7 [167.1 to 222.1] | 190.5 [171.3 to 211.8] | 199.2 [172.6 to 229.8] | 200.9 [168.2 to 239.9] | 199.3 [180.0 to 220.7] | 137.1 [118.3 to 158.8] | 168.9 [144.1 to 197.8]
  Day 182 (B/Phuket/3073/2013 (Yamagata Lineage)) | 132.2 [115.3 to 151.6] | 126.8 [115.1 to 139.6] | 127.2 [111.6 to 144.8] | 143.4 [121.8 to 168.8] | 131.4 [119.3 to 144.7] | 111.2 [98.4 to 125.8] | 125.3 [107.8 to 141.1]
  Day 0 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 69.9 [62.9 to 77.7] | 75.8 [70.0 to 82.1] | 70.3 [62.6 to 78.8] | 77.7 [69.4 to 87.1] | 71.8 [66.5 to 77.6] | 73.0 [65.6 to 81.2] | 71.3 [64.3 to 79.0]
  Day 28 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 140.1 [120.8 to 162.6] | 147.9 [133.9 to 163.3] | 128.8 [112.2 to 147.9] | 140.7 [121.3 to 163.0] | 122.1 [110.4 to 135.1] | 141.7 [122.0 to 164.7] | 149.2 [127.8 to 174.2]
  Day 56 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 132.0 [113.0 to 154.1] | 132.2 [119.1 to 146.8] | 126.4 [107.8 to 140.8] | 120.5 [103.1 to 140.8] | 150.4 [134.5 to 168.2] | 125.4 [107.5 to 146.3] | 119.3 [101.0 to 141.0]
  Day 182 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 87.1 [73.9 to 102.6] | 90.2 [81.0 to 100.4] | 91.4 [77.2 to 108.3] | 85.1 [71.8 to 101.0] | 97.8 [87.4 to 109.5] | 86.1 [74.2 to 100.0] | 84.0 [71.2 to 99.1]

5. Secondary Outcome: HAI Titers Specific for Vaccine-homologous A and B Influenza Strains Expressed as Geometric Mean Fold Ratio (GMFR)
Description: HAI antibody titers specific for the HA receptor binding domains of vaccine-homologous A and B strain(s) expressed as GMFR on Day 28,56 and 182.
Time Frame: Day 28 - Day 182
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Ratio
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 149 | 295 | 147 | 121 | 290 | 143 | 144
Fold Ratio
  Day 28 (A/Michigan/45/2015 (H1N1)) | 1.9 [1.7 to 2.1] | 1.7 [1.6 to 1.9] | 1.7 [1.6 to 2.0] | 1.5 [1.4 to 1.7] | 1.7 [1.6 to 1.9] | 1.9 [1.7 to 2.2] | 1.8 [1.6 to 2.1]
  Day 56 (A/Michigan/45/2015 (H1N1)) | 1.6 [1.4 to 1.8] | 1.4 [1.3 to 1.5] | 1.4 [1.3 to 1.6] | 1.2 [1.1 to 1.4] | 1.8 [1.6 to 1.9] | 1.5 [1.3 to 1.7] | 1.4 [1.2 to 1.6]
  Day 182 (A/Michigan/45/2015 (H1N1)) | 1.3 [1.2 to 1.5] | 1.2 [1.1 to 1.3] | 1.3 [1.2 to 1.5] | 1.1 [1.0 to 1.3] | 1.4 [1.3 to 1.6] | 1.4 [1.3 to 1.5] | 1.3 [1.1 to 1.4]
  Day 28 (B/Colorado/06/2017 (Victoria Lineage)) | 1.6 [1.4 to 1.8] | 1.6 [1.5 to 1.7] | 1.6 [1.5 to 1.8] | 1.6 [1.4 to 1.8] | 1.4 [1.3 to 1.4] | 1.9 [1.6 to 2.1] | 1.6 [1.4 to 1.8]
  Day 56 (B/Colorado/06/2017 (Victoria Lineage)) | 1.3 [1.2 to 1.5] | 1.4 [1.3 to 1.5] | 1.4 [1.2 to 1.6] | 1.4 [1.2 to 1.6] | 1.6 [1.5 to 1.7] | 1.6 [1.4 to 1.8] | 1.3 [1.2 to 1.4]
  Day 182 (B/Colorado/06/2017 (Victoria Lineage)) | 1.2 [1.1 to 1.3] | 1.2 [1.1 to 1.3] | 1.3 [1.2 to 1.4] | 1.2 [1.1 to 1.4] | 1.4 [1.3 to 1.5] | 1.4 [1.3 to 1.6] | 1.2 [1.1 to 1.3]
  Day 28 (B/Phuket/3073/2013 (Yamagata Lineage)) | 1.9 [1.7 to 2.2] | 2.0 [1.9 to 2.2] | 2.2 [1.9 to 2.5] | 2.0 [1.7 to 2.4] | 1.8 [1.7 to 2.0] | 1.4 [1.3 to 1.5] | 2.0 [1.8 to 2.3]
  Day 56 (B/Phuket/3073/2013 (Yamagata Lineage)) | 1.9 [1.7 to 2.1] | 2.0 [1.8 to 2.1] | 2.1 [1.8 to 2.4] | 1.9 [1.7 to 2.3] | 2.0 [1.8 to 2.2] | 1.4 [1.3 to 1.5] | 2.0 [1.7 to 2.3]
  Day 182 (B/Phuket/3073/2013 (Yamagata Lineage)) | 1.3 [1.2 to 1.4] | 1.3 [1.2 to 1.4] | 1.4 [1.2 to 1.5] | 1.4 [1.2 to 1.6] | 1.3 [1.2 to 1.4] | 1.1 [1.0 to 1.2] | 1.4 [1.3 to 1.6]
  Day 28 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 2.0 [1.8 to 2.3] | 2.0 [1.8 to 2.1] | 1.8 [1.6 to 2.0] | 1.8 [1.6 to 2.1] | 1.7 [1.6 to 1.8] | 1.9 [1.7 to 2.2] | 2.1 [1.8 to 2.4]
  Day 56 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 1.9 [1.6 to 2.2] | 1.7 [1.6 to 1.9] | 1.8 [1.6 to 2.1] | 1.6 [1.4 to 1.8] | 2.1 [1.9 to 2.3] | 1.7 [1.5 to 2.0] | 1.7 [1.4 to 2.0]
  Day 182 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 1.2 [1.1 to 1.4] | 1.2 [1.1 to 1.3] | 1.3 [1.1 to 1.5] | 1.1 [1.0 to 1.3] | 1.4 [1.3 to 1.5] | 1.2 [1.0 to 1.3] | 1.2 [1.0 to 1.4]

6. Secondary Outcome: Number of Participants Who Seroconverted as Determined by HAI Titers Specific for Vaccine-homologous A and B Influenza Strains
Description: HAI antibody titers specific for the HA receptor binding domains of vaccine-homologous A and B strain(s) expressed as SCR on Day 28,56 and 182.
Time Frame: Day 28 - Day 182
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 149 | 295 | 147 | 121 | 290 | 143 | 144
Participants
  Day 28 (A/Michigan/45/2015 (H1N1)) | 31 | 41 | 22 | 13 | 52 | 32 | 26
  Day 56 (A/Michigan/45/2015 (H1N1)) | 15 | 23 | 10 | 4 | 39 | 10 | 13
  Day 182 (A/Michigan/45/2015 (H1N1)) | 8 | 14 | 7 | 5 | 23 | 8 | 6
  Day 28 (B/Colorado/06/2017 (Victoria Lineage)) | 25 | 32 | 20 | 20 | 23 | 32 | 18
  Day 56 (B/Colorado/06/2017 (Victoria Lineage)) | 6 | 21 | 7 | 8 | 21 | 12 | 8
  Day 182 (B/Colorado/06/2017 (Victoria Lineage)) | 7 | 11 | 7 | 7 | 12 | 9 | 6
  Day 28 (B/Phuket/3073/2013 (Yamagata Lineage)) | 32 | 70 | 43 | 35 | 57 | 10 | 37
  Day 56 (B/Phuket/3073/2013 (Yamagata Lineage)) | 24 | 46 | 33 | 27 | 52 | 7 | 34
  Day 182 (B/Phuket/3073/2013 (Yamagata Lineage)) | 6 | 11 | 7 | 10 | 10 | 0 | 5
  Day 28 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 40 | 68 | 29 | 23 | 54 | 31 | 37
  Day 56 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 29 | 41 | 16 | 11 | 52 | 21 | 20
  Day 182 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 16 | 10 | 10 | 5 | 17 | 6 | 15

7. Secondary Outcome: Number of Participants Who Had Seroprotection as Determined by HAI Titers Specific for Vaccine-homologous A and B Influenza Strains
Description: HAI antibody titers specific for the HA receptor binding domains of vaccine-homologous A and B strain(s) expressed as SPR on Day 28,56 and 182.
Time Frame: Day 28 - Day 182
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 149 | 295 | 147 | 121 | 290 | 143 | 144
participants
  Day 28 (A/Michigan/45/2015 (H1N1)) | 133 | 260 | 131 | 105 | 257 | 133 | 126
  Day 56 (A/Michigan/45/2015 (H1N1)) | 94 | 174 | 92 | 58 | 203 | 95 | 76
  Day 182 (A/Michigan/45/2015 (H1N1)) | 106 | 188 | 99 | 73 | 212 | 110 | 88
  Day 28 (B/Colorado/06/2017 (Victoria Lineage)) | 149 | 295 | 147 | 120 | 290 | 142 | 144
  Day 56 (B/Colorado/06/2017 (Victoria Lineage)) | 141 | 282 | 139 | 114 | 282 | 134 | 129
  Day 182 (B/Colorado/06/2017 (Victoria Lineage)) | 141 | 277 | 136 | 115 | 280 | 140 | 134
  Day 28 (B/Phuket/3073/2013 (Yamagata Lineage)) | 149 | 295 | 147 | 120 | 290 | 143 | 143
  Day 56 (B/Phuket/3073/2013 (Yamagata Lineage)) | 146 | 292 | 141 | 118 | 286 | 137 | 135
  Day 182 (B/Phuket/3073/2013 (Yamagata Lineage)) | 137 | 279 | 133 | 114 | 274 | 134 | 130
  Day 28 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 147 | 293 | 145 | 120 | 285 | 142 | 143
  Day 56 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 130 | 272 | 126 | 105 | 265 | 124 | 120
  Day 182 (A/Singapore/INFIMH-16-0019/2016 (H3N2)) | 109 | 233 | 108 | 88 | 224 | 113 | 104

8. Secondary Outcome: HAI Titers Specific for Antigenically-drifted Influenza Strains Expressed as GMT
Description: HAI antibody titers specific for antigenically-drifted influenza strains, at Days 0,28, 56 and 182 expressed as geometric man titer (GMT).
Time Frame: Day 0 - Day 182
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: titers
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 149 | 295 | 147 | 121 | 290 | 143 | 144
titers
  Day 0 (A/Switzerland/9715293/2013 (H3N2)) | 51.7 [46.0 to 58.1] | 53.8 [49.1 to 58.9] | 57.1 [50.1 to 65.1] | 55.3 [48.3 to 63.3] | 55.7 [51.1 to 60.7] | 60.5 [53.4 to 68.6] | 54.3 [47.6 to 61.9]
  Day 28 (A/Switzerland/9715293/2013 (H3N2)) | 118.5 [101.0 to 139.1] | 124.7 [112.7 to 138.1] | 120.0 [103.4 to 139.2] | 115.1 [97.3 to 136.1] | 105.4 [95.1 to 116.9] | 102.7 [86.7 to 121.6] | 138.2 [115.7 to 165.0]
  Day 56 (A/Switzerland/9715293/2013 (H3N2)) | 93.9 [81.0 to 108.0] | 91.4 [83.1 to 100.5] | 92.2 [80.4 to 105.7] | 88.3 [75.3 to 103.6] | 97.3 [87.7 to 108.0] | 77.2 [66.2 to 89.9] | 96.3 [81.3 to 114.0]
  Day 182 (A/Switzerland/9715293/2013 (H3N2)) | 73.4 [63.8 to 84.5] | 72.4 [66.1 to 79.2] | 73.4 [64.1 to 84.0] | 72.0 [62.3 to 83.0] | 77.2 [69.8 to 85.4] | 66.1 [57.3 to 76.4] | 77.2 [66.6 to 86.6]

9. Secondary Outcome: HAI Titer Responses Specific for Antigenically-drifted Influenza Strains Expressed as GMFR
Description: HAI antibody titer responses specific for antigenically-drifted influenza strains, at Days 28, 56, and 182 expressed as Geometric Fold Ratio.
Time Frame: Day 28 - Day 182
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Fold Ratio
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 149 | 295 | 147 | 121 | 290 | 143 | 144
Fold Ratio
  Day 28 (A/Switzerland/9715293/2013 (H3N2)) | 2.3 [2.0 to 2.6] | 2.3 [2.1 to 2.5] | 2.1 [1.9 to 2.4] | 2.1 [1.8 to 2.4] | 1.9 [1.7 to 2.1] | 1.7 [1.5 to 1.9] | 2.5 [2.2 to 3.0]
  Day 56 (A/Switzerland/9715293/2013 (H3N2)) | 1.8 [1.6 to 2.1] | 1.7 [1.5 to 1.9] | 1.6 [1.4 to 1.8] | 1.6 [1.4 to 1.8] | 1.7 [1.6 to 1.9] | 1.3 [1.1 to 1.4] | 1.8 [1.5 to 2.1]
  Day 182 (A/Switzerland/9715293/2013 (H3N2)) | 1.4 [1.3 to 1.6] | 1.3 [1.2 to 1.4] | 1.3 [1.2 to 1.4] | 1.3 [1.2 to 1.5] | 1.4 [1.3 to 1.5] | 1.1 [1.0 to 1.2] | 1.4 [1.3 to 1.6]
  Day 28 (A/Wisconsin/19/2017 (H3N2)) | 2.4 [2.0 to 2.8] | 2.5 [2.3 to 2.8] | 2.3 [2.0 to 2.6] | 2.1 [1.8 to 2.5] | 1.9 [1.8 to 2.2] | 2.4 [2.1 to 2.8] | 2.7 [2.2 to 3.2]
  Day 56 (A/Wisconsin/19/2017 (H3N2)) | 2.0 [1.7 to 2.3] | 1.9 [1.7 to 2.1] | 1.9 [1.7 to 2.2] | 1.7 [1.4 to 2.0] | 2.4 [2.2 to 2.7] | 1.8 [1.6 to 2.1] | 1.9 [1.6 to 2.2]
  Day 182 (A/Wisconsin/19/2017 (H3N2)) | 1.4 [1.2 to 1.6] | 1.3 [1.2 to 1.4] | 1.4 [1.3 to 1.6] | 1.3 [1.1 to 1.5] | 1.5 [1.4 to 1.6] | 1.3 [1.1 to 1.4] | 1.3 [1.1 to 1.4]

10. Secondary Outcome: Number of Participants Who Seroconverted as Determined by HAI Titers Specific for Antigenically-drifted Influenza Strains
Description: HAI antibody titers specific for antigenically-drifted influenza strains, at Days 28, 56 and 182 expressed as SCR.
Time Frame: Day 28 - Day 182
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 149 | 295 | 147 | 121 | 290 | 143 | 144
participants
  Day 28 (A/Switzerland/9715293/2013 (H3N2)) | 45 | 89 | 38 | 28 | 63 | 20 | 47
  Day 56 (A/Switzerland/9715293/2013 (H3N2)) | 15 | 27 | 9 | 8 | 26 | 5 | 18
  Day 182 (A/Switzerland/9715293/2013 (H3N2)) | 15 | 22 | 6 | 9 | 21 | 4 | 14
  Day 28 (A/Wisconsin/19/2017 (H3N2)) | 50 | 94 | 41 | 30 | 69 | 44 | 50
  Day 56 (A/Wisconsin/19/2017 (H3N2)) | 28 | 49 | 23 | 16 | 63 | 18 | 26
  Day 182 (A/Wisconsin/19/2017 (H3N2)) | 8 | 17 | 8 | 8 | 21 | 6 | 8

11. Secondary Outcome: Number of Participants Who Had Seroprotection as Determined by HAI Titers of Antigenically-drifted Influenza Strains
Description: HAI antibody titers specific for antigenically-drifted influenza strains, at Days 28, 56 and 182 expressed as SPR.
Time Frame: Day 28 - Day 182
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine
Number analyzed (Participants) | 149 | 295 | 147 | 121 | 290 | 143 | 144
participants
  Day 28 (A/Switzerland/9715293/2013 (H3N2)) | 139 | 288 | 138 | 112 | 276 | 129 | 135
  Day 56 (A/Switzerland/9715293/2013 (H3N2)) | 107 | 215 | 108 | 85 | 212 | 87 | 101
  Day 182 (A/Switzerland/9715293/2013 (H3N2)) | 113 | 234 | 112 | 90 | 224 | 101 | 112
  Day 28 (A/Wisconsin/19/2017 (H3N2)) | 130 | 276 | 134 | 108 | 246 | 129 | 130
  Day 56 (A/Wisconsin/19/2017 (H3N2)) | 110 | 233 | 111 | 87 | 245 | 109 | 103
  Day 182 (A/Wisconsin/19/2017 (H3N2)) | 104 | 215 | 103 | 91 | 213 | 105 | 105

ADVERSE EVENTS:
Time Frame: 6 Months
Description: Serious Adverse Events, Other (Not Including Serious) Adverse Events
Arm/Group | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose A | Quad-NIV Preformulated With Adjuvant Dose B | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A | Quad-NIV Without Adjuvant | Licensed High-Dose Trivalent Influenza Vaccine | Licensed Quadrivalent Influenza Vaccine
All-Cause Mortality (participants affected / at risk) | 1/157 | 3/305 | 0/156 | 2/132 | 0/311 | 0/153 | 1/151
Serious Adverse Events (participants affected / at risk) | 12/157 | 21/305 | 16/156 | 22/132 | 7/311 | 8/153 | 6/151
Other Adverse Events (participants affected / at risk) | 4/157 | 14/305 | 7/156 | 2/132 | 16/311 | 10/153 | 2/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A (N=157) | Quad-NIV Preformulated With Adjuvant Dose A (N=305) | Quad-NIV Preformulated With Adjuvant Dose B (N=156) | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A (N=132) | Quad-NIV Without Adjuvant (N=311) | Licensed High-Dose Trivalent Influenza Vaccine (N=153) | Licensed Quadrivalent Influenza Vaccine (N=151)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroptosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quad-NIV Bedside Mix of Antigen and Adjuvant Dose A (N=157) | Quad-NIV Preformulated With Adjuvant Dose A (N=305) | Quad-NIV Preformulated With Adjuvant Dose B (N=156) | Quad-NIV Preformulated With Increased B HA Adjuvant Dose A (N=132) | Quad-NIV Without Adjuvant (N=311) | Licensed High-Dose Trivalent Influenza Vaccine (N=153) | Licensed Quadrivalent Influenza Vaccine (N=151)
Blood urea increased (Investigations) | 4 (4) | 14 (14) | 7 (7) | 2 (2) | 16 (16) | 10 (10) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was terminated at 182 days after initial dosing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT03658629/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/29/NCT03658629/SAP_001.pdf